CLINICAL TRIAL: NCT00645359
Title: Pilot Study of Diffusion MRI as a Tool for Early Evaluation of Tumor Response in Diffuse Large B Cell Lymphoma
Brief Title: Pilot Study of dMRI as a Tool for Early Evaluation of Tumor Response in Diffuse Large B-cell Lymphoma
Acronym: dMRI
Status: Terminated | Type: Observational
Why Stopped: Insufficient resources to evaluate pilot, second to shift in research priorities
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2006.063; HUM 6946 (Other: University of Michigan Medical School IRB)
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: dMRI; diffusion MRI; Diffuse large B-cell lymphoma; DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diffusion MRI: Patients will undergo a Diffusion MRI (dMRI) at baseline and 7 days.
  Interventions: Procedure: diffusion MRI

INTERVENTIONS:
Procedure: diffusion MRI — Diffusion MRI involves using MRI scanning to measure water transport at the cellular level. In this study, dMRI is being used to measure the response of tumors to chemotherapy.
  Other Names: dMRI, diffusion MRI, diffusion Magnetic Resonance Imaging

SUMMARY:
This research study is designed to test whether the results of a diffusion MRI scan performed after one cycle of chemotherapy for lymphoma can accurately predict the outcome of treatment for individual patients.

DETAILED DESCRIPTION:
Different types of functional imaging are under investigation as a tool to predict response to treatment, as imaging soon after starting therapy might be able to better define the likelihood of response. Functional imaging refers to scans that measure characteristics other than size and shape (anatomic imaging), as measured by CT scans. We are interested in evaluating the potential value of diffusion Magnetic Resonance Imaging (dMRI), which in some settings can be used very early in treatment in predicting patients' response to treatment.

Diffusion MRI (dMRI) detects changes in cell structure, and has the potential to detect and measure cell changes that occur in response to treatment. Several groups are investigating the use of dMRI to monitor treatment responses. This strategy has been most frequently explored in humans in patients with brain tumors, where dMRI has been demonstrated to predict response to treatment early after starting treatment. A few studies have looked at response in other cancers. These studies showed early changes in patients who later responded to treatment, with changes seen within one to 2 weeks.

Although diffusion MRI has been shown to be useful in several cancer types, it has not been explored in the evaluation of lymphoma. This pilot study will evaluate the imaging characteristics of Diffuse Large B-Cell Lymphoma (DLBCL) by dMRI prior to treatment and 7 days after initial chemotherapy in order to explore whether dMRI is useful in evaluating the response of lymphoma to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new diagnosis of CD20 Positive diffuse large B cell lymphoma (LBCL) of any stage, including subtypes mediastinal large B cell, centroblastic, immunoblastic, T cell rich B cell and anaplastic B cell lymphoma, who will receive standard R/CHOP as first line chemotherapy will be included.
* Patients must be age 18 or older.
* No selection will be made on the basis of gender, race or ethnicity.

Exclusion Criteria:

* Patients will be excluded if the diagnosis of diffuse large B cell lymphoma cannot be confirmed.
* Patients receiving treatment other than R/CHOP or R/CHOP followed by radiotherapy or who have previously been treated for DLBCL will be excluded. - Patients with HIV infection will also be excluded. No selection will be made based on other medical problems or laboratory values, except as they affect the patient's eligibility to receive standard R/CHOP chemotherapy as determined by the treating physician.
* Patients who have magnetic metal implants or fragments in their body that are incompatible with MRI will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lymphoma of any stage or subtype (including all Hodgkin's and non-Hodgkin's lymphomas), previously untreated or in relapse, who are starting on a new line of therapy with intent to induce a remission.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2006-11; Primary Completion 2011-07 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Diffusion MRI: Participants will undergo two Diffusion MRIs (Magnetic Resonance Imaging) at at baseline and Cycle 1 Day 8.
Period: Overall Study
Arm/Group | Diffusion MRI
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diffusion MRI
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 61 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Apparent Diffusion Coefficient
Description: To assess whether changes in the apparent diffusion coefficient (ADC) during the early phase of chemotherapy are detectable in lymphoma, the ADC value will be calculated at the voxel level, on baseline and Day 8, and the mean difference will be calculated.
Time Frame: Baseline and Day 8
Population: No patients were analyzed due to insufficient resources, secondary to shifting research priorities.
Arm/Group | Diffusion MRI
Number analyzed (Participants) | 0

2. Primary Outcome: The Odds Ratio (OR) Between Tumor Response (Based on Changes in MR Imaging) and Duration of Response
Description: To correlate the changes on MR images with the tumor response after completion of chemotherapy and duration of response. Tumor response will be determined by the clinical evaluation, tumor dimensions, and metabolic response as assessed by 18-Fluoro-deoxy.
Time Frame: 2 years
Population: No patients were analyzed due to insufficient resources, secondary to shifting research priorities.
Arm/Group | Diffusion MRI
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Only events related to the Diffusion MRI were reportable.
Arm/Group | Diffusion MRI
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
This study was not completed due to insufficient resources to evaluate the pilot phase of the study, secondary to shifting research priorities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes